CLINICAL TRIAL: NCT07074600
Title: Clinical Efficacy of Electroacupuncture Therapy on Limb Dysfunction in Ischemic Stroke Patients at High-Altitude Regions: A Multi-center Randomized Double-blind Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiyang Zheng (Other)
Collaborators: Qinghai People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Kaiyang Zheng, student, Qinghai University
Organization: Qinghai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PJ202501-23
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Limb Dysfunction in Ischemic Stroke Patients at High-Altitude Regions
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture Therapy (Experimental): Participants will be randomized into an experimental group and a control group. The experimental group will receive daily electroacupuncture therapy for a standardized 14-day course, with comprehensive functional and neurological assessments conducted at pre-intervention (baseline) and post-intervention timepoints. The control group will undergo daily sham acupuncture under identical conditions, including matching treatment duration and assessment schedules. Electroacupuncture administration will target acupoints spanning cranial, upper limb, and lower limb anatomical domains.
  Interventions: Device: Electroacupuncture Therapy
- Sham electroacupuncture intervention (Experimental): Participants in the control group will receive daily sham electroacupuncture therapy over a standardized 14-day therapeutic course. Comprehensive functional and neurological assessments will be conducted at pre-intervention (baseline) and post-intervention timepoints. Sham electroacupuncture procedures will target non-acupoint locations outside recognized cranial, upper limb, and lower limb anatomical domains.
  Interventions: Device: Sham electroacupuncture intervention

INTERVENTIONS:
Device: Electroacupuncture Therapy — Participants in the experimental group will receive daily electroacupuncture therapy over a standardized 14-day therapeutic course. Comprehensive functional and neurological assessments will be conducted at pre-intervention (baseline) and post-intervention timepoints. Acupoint selection will target anatomical domains spanning the cranial, upper limb, and lower limb regions.
  Other Names: Electroacupuncture
  Arms: Electroacupuncture Therapy
Device: Sham electroacupuncture intervention — Participants in the control group will receive daily sham electroacupuncture therapy over a standardized 14-day therapeutic course. Comprehensive functional and neurological assessments will be conducted at pre-intervention (baseline) and post-intervention timepoints. Sham electroacupuncture procedures will target non-acupoint locations outside recognized cranial, upper limb, and lower limb anatomical domains.
  Other Names: Sham electroacupuncture
  Arms: Sham electroacupuncture intervention

SUMMARY:
The purpose of this clinical trial is to investigate the efficacy of electroacupuncture therapy for limb dysfunction in ischemic stroke patients residing at high-altitude regions. This study aims to address the following research questions: 1. Whether electroacupuncture therapy demonstrates clinical effectiveness in managing limb dysfunction among ischemic stroke patients in high-altitude regions. 2. Whether electroacupuncture therapy maintains an acceptable safety profile in this specific population.

Researchers will conduct a comparative analysis between the active electroacupuncture intervention group and a sham-electroacupuncture control group to evaluate therapeutic efficacy. Participants will: 1. Undergo daily electroacupuncture treatment sessions for a standardized 14-day therapeutic course. 2. Complete comprehensive functional assessments and neurological evaluations at baseline and post-intervention timepoints.

ELIGIBILITY:
Inclusion Criteria:

* (1) Meeting diagnostic criteria for ischemic stroke ; (2) Aged 18-75 years ; (3) Total stroke episodes < 3 ; (4) Current stroke with disease course of 2 weeks to 3 months ; (5) Severity of limb motor impairment assessed by the National Institutes of Health Stroke Scale (NIHSS) score .

Exclusion Criteria:

* (1) Patients with transient ischemic attack (TIA), cerebral hemorrhage, or reversible ischemic neurological deficit (RIND); (2) Patients with intracranial space-occupying lesions; (3) Patients with severe aphasia or other complications impairing scale assessment compliance; (4) Pregnant or lactating women, or those planning pregnancy; (5) Patients with acupuncture contraindications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Scale (FMA) | "Baseline"，"Day 7"，"Day 14"
Fugl-Meyer Assessment Scale (FMA) | "Baseline"，"Day 7"，"Day 14"
  Assessments were conducted at baseline (pre-intervention), day 7 of treatment, and post-intervention. The evaluation comprises 33 items for upper extremity motor function and 17 items for lower extremity motor function. Each item is scored 2 points for full completion, 1 point for partial completion, and 0 points for inability to complete. The total score ranges from 0 to 66 for upper extremities and 0 to 34 for lower extremities, with higher scores indicating better motor function.

SECONDARY OUTCOMES:
Activities of Daily Living Assessment Scale (ADL) Score | "Baseline"，"Day 7"，"Day 14"
  Assessments were conducted at baseline (pre-intervention), day 10 of treatment, and post-intervention. The ADL assessment scale is primarily used to evaluate the activities of daily living and functional status in stroke patients, encompassing 11 items related to 10 fundamental aspects of self-care and mobility. Each item is scored on a scale of 0 to 15 points, with the sum of all items constituting the ADL score. Higher scores indicate better daily living ability.

IPD SHARING:
Plan to Share IPD: No